CLINICAL TRIAL: NCT02578173
Title: Evaluation of a Novel Method of Contrast Volume Quantification - AVERT PLUS 2.0
Status: Completed | Type: Observational
Sponsor: Anand Prasad (Other)
Responsible Party: Sponsor-Investigator, Anand Prasad, Assistant Professor of Medicine, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Other Study IDs: HSC20150682H
Record Dates: First submitted 2015-10-10; First posted 2015-10-16 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AVERT PLUS: The AVERT PLUS will be used on the first 10 patients enrolled in the study. The AVERT PLUS is a contrast monitoring system which is used to precisely measure the volume of contrast delivered to the patient.
  Interventions: Device: AVERT PLUS
- Non device group: The second group of 10 patients will undergo the scheduled angiography using the standard method of measuring contrast dye delivery.

INTERVENTIONS:
Device: AVERT PLUS
  Groups: AVERT PLUS

SUMMARY:
Purpose: To evaluate the accuracy of the AVERT PLUS to monitor contrast volume used during angiographic procedures. This will be a first in man prospective observational study of the accuracy of this system to quantify contrast volume used during clinically indicated angiography in the cardiac catheterization laboratory.

DETAILED DESCRIPTION:
Research Design:

The AVERT PLUS is an FDA 510K cleared device which consists of 1) a contrast delivery modulator designed to reduce unnecessary contract dye delivery to the patient during angiography (coronary or peripheral) and 2) a concomitant contrast monitoring system to precisely measure contrast volume delivered to the patient. This will be a first in man prospective observational study of the accuracy of this system to quantify contrast volume used during clinically indicated angiography in the cardiac catheterization laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing clinically indicated coronary or peripheral angiography

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiovascular disease who are undergoing clinically indicated coronary or peripheral angiography
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Observational study of the accuracy of the AVERT PLUS CM system to quantify contrast volume during a clinically indicated procedure. | The total volume of contrast received by the subject will be measured at the conclusion of the angiography procedure, procedure duration from 30 minutes to 4 hours dependent on patient's clinical status; no further measurements thereafter.
  The fluid volume of contrast media used during the angiography procedure will be measured in milliliters.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Shepard, Study Director — Osprey Medical, Inc